CLINICAL TRIAL: NCT00594971
Title: A Shared Care Approach for Seriously Ill Cancer Patients Between General Practice, Discharge Department and a Specialist Palliative Care Team
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems has forced us to change the design of this study from a clinical trial to a comparative study of 3 different groups of patients.
Sponsor: University of Aarhus (Other)
Collaborators: Research Unit for General Practice, Aarhus University (Other); Aarhus University Hospital (Other)
Responsible Party: Professor Frede Olesen, Research Unit for General Practice, Aarhus University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 15273887; ISRCTN15273887
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Palliative Care; Neoplasms
Keywords: Health Services Research; Family practice
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- B (Other): 90 terminally ill cancer patients will be referred to a specialist palliative care team at time of discharge.
  Interventions: Other: Referral to a specialist palliative care team.
- C (Other): 90 terminally ill cancer patients will be discharged from hospital with extra effort put into improving the communication between the hospital and the primary sector.
  Interventions: Other: Organisational intervention
- A (No Intervention): 90 terminally ill cancer patients will be discharged from hospital, receiving usual care.

INTERVENTIONS:
Other: Organisational intervention — A shared care approach in which extra effort is put into improving the communication between the hospital and the primary sector.
  Arms: C
Other: Referral to a specialist palliative care team. — Discharge with referral to a specialist palliative care team. This is a patient-centred shared care model in which the palliative team helps to organise the patient's treatment and care.
  Arms: B

SUMMARY:
Background:

Approximately one third of all deaths in Denmark are caused by cancer. Both Danish and international research shows that the majority of terminally ill cancer patients wish to die at home. In Denmark only about 25% has this wish fulfilled. The General Practitioner (GP) has traditionally had the full responsibility for the palliative care of terminally ill cancer patients. In recent years changes have been made to the organisation of palliative care: some hospitals have set up specialised palliative care teams and in some areas of Denmark hospices have been established.

Recent research defines a problem when it comes to communication between the hospital and general practice when the patient is being discharged. This is often done in a way that can cause the patient to feel "left in limbo", especially if it is not completely clear to the patient and his or her relatives who has the responsibility for the palliative care.

Objective:

1. To describe consequences for patients, relatives and health care professionals of three different ways of organising palliative care
2. To collect data which describes patients who are candidates to a shared care approach between general practice and a specialised palliative care team
3. To collect data which describes the palliative phase (place of death and palliative care, admissions to hospital, involvement of GP and district nurse etc.)
4. To describe terminally ill cancer patients and their relatives expectations of the health care system

270 terminally ill cancer patients will be invited to take part in the study. Data will be collected by interview with patients and questionnaires for patients, relatives and involved health care professionals.

DETAILED DESCRIPTION:
The intervention in the study is of organisational character. The patients will be randomised into two groups (groups B and C). A group of usual care patients will be included primary to the intervention (group A). The groups are:

A. Usual discharge with regular discharge letter to the GP. The GP, together with the community nurse, is responsible for the palliative care, including referral to a specialist palliative care team, hospice, hospital, etc., if necessary

B. Discharge with referral to a specialist palliative care team. This is a patient-centred shared care model in which the palliative team helps to organise the patient's treatment and care

C. Discharge with extra effort put into improving the communication between the hospital and the GP. The GP will receive a phone call from the doctor who is discharging the patient, a detailed discharge letter, written information about the patient's type of cancer and acute oncological symptoms, name and phone number of the community nurse and name and phone number of a specialist in palliative medicine, who can be contacted for advice. This is a shared care model, where focus is on supporting the health care professionals.

ELIGIBILITY:
Inclusion Criteria:

In order to be included the patients have to be diagnosed as suffering from terminal cancer. The patients should also:

1. Be 18 years or older
2. Be able to speak and write Danish fluently
3. Give written and spoken consent
4. Be able to manage in their own home, with or without the help of carers and district nurses
5. Be informed about the diagnosis, also that it is incurable
6. Be registered as suffering from a terminal illness or fulfil the criteria for this -

Exclusion Criteria:

Patients are excluded if they:

1. Have a low level of cognitive skills, which makes it difficult for them to fill in a questionnaire
2. Are residents of a nursing home at the time of inclusion
3. Are receiving oncologic treatment which requires attending an out-patients clinic regularly
4. Already have established contact with a specialist palliative care team at the time of inclusion -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-10 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Patients wish for place of death and place of terminal care fulfilled | The patient will be asked about preference for place of death and place for terminal care at inclusion and a month later. At the time of death we will be able to establish weather the patient had his or her wishes fulfilled.
Relative amount of time spent in hospital in the terminal phase | At the patients time of death we will be able to count number of days spent in hospital using the hospitals electronic patient files.
A subjective measure of the patients symptoms and quality of life (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire of Palliative care [EORTC-QLQ-15-PAL]) | Will be measured at the time of inclusion and a month later.

SECONDARY OUTCOMES:
Patient's satisfaction regarding the services of the GP, district nurse and local hospital | Will be measured at inclusion and one month later.
Patient's experiences regarding cooperation and information sharing in the health care system. | Will be measured at inclusion and one month later.
Relative's satisfaction regarding the services of the GP, district nurse and local hospital. | Will be measured at inclusion, one month later and 2 months after the patients death.
Relative's experiences regarding cooperation and information sharing in the health care system. | Will be measured at inclusion, one month later and 2 months after the patients death.
Relative's experiences regarding the palliative treatment of the patient. | Will be measured at inclusion, one month later and 2 months after the patients death.
Subjective burden of relative (Burden Scale for Family Caregivers [BSFC]). | Will be measured at inclusion and one month later.
GPs evaluation of the terminal phase. | Will be measured after the patients death.
District nurses evaluation of the terminal phase. | Will be measured after the patients death.
Hospital doctors evaluation of the terminal phase. | Will be measured after the patients death.

CONTACTS AND LOCATIONS:
Overall Officials: Frede Olesen, Professor, Study Director — Research Unit for General Practice, Aarhus University